CLINICAL TRIAL: NCT03895099
Title: Feasibility and Efficacy of a New Ovarian Stimulation Regimen With RANDom Start, Use of Corifollitropin Alpha and Progestin Protocol for Oocyte donorS
Brief Title: New Ovarian Stimulation With Random Start, Use of Progestin Protocol for Oocyte Donors
Acronym: RANDOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RANDOS
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A - Early follicular phase (Experimental): Treatment by desogestrel at day 1 to day 3
  Interventions: Drug: Desogestrel early follicular phase
- B - Medium follicular phase (Experimental): Treatment by desogestrel at day 4 to day 7
  Interventions: Drug: Desogestrel medium follicular phase
- C - Late follicular phase (Experimental): Treatment by desogestrel at day 7 to day 11
  Interventions: Drug: Desogestrel ovulatory phase
- D - Ovulatory Phase (Experimental): Treatment by desogestrel at day 12 to day 15
  Interventions: Drug: Desogestrel late follicular phase
- E - Luteal phase (Experimental): Treatment by desogestrel at day 16 to day 30
  Interventions: Drug: Desogestrel luteal phase

INTERVENTIONS:
Drug: Desogestrel early follicular phase — Start of ovarian stimulation in early follicular phase
  Arms: A - Early follicular phase
Drug: Desogestrel medium follicular phase — Start of ovarian stimulation in medium follicular phase
  Arms: B - Medium follicular phase
Drug: Desogestrel ovulatory phase — Start of ovarian stimulation in ate follicular phase
  Arms: C - Late follicular phase
Drug: Desogestrel late follicular phase — Start of ovarian stimulation in ovulatory Phase
  Arms: D - Ovulatory Phase
Drug: Desogestrel luteal phase — Start of ovarian stimulation in luteal phase
  Arms: E - Luteal phase

SUMMARY:
Oocyte donation is a cumbersome and demanding procedure, involving an injectable hormonal treatment for an average duration of 12 days, according to the protocols, 1 to several daily injections. The objective of this study is to show that treatments can be simplified without reducing the number of oocytes that have been punctured, by blocking the luteinizing hormone (LH) surge by using oral progesterone and by limiting the number of injections of gonadotropins using corifollitropin alpha, regardless of the start date of the pacing protocol during a natural cycle.

DETAILED DESCRIPTION:
Medically assisted procreation can help infertile patients with a panel of techniques adapted to various causes of infertility. In most cases, these techniques use patients' own gametes. However, despite the medical advances, it is still impossible today to regenerate gametic cells when they have disappeared from the gonads. Especially for women with premature ovarian failure, the only feasible option is to receive oocytes from a third-party donor. In France, the principle of free and anonymous applies to the donation and no compensation is allowed outside the reimbursement of expenses incurred. Oocyte donors are women volunteers who agree to undergo heavy medical treatment to help other women, without any other consideration so that the recognition of their donation. It is important for these women to minimize the risks involved, to simplify and minimize ovarian stimulation treatments, which are generally injections and to offer maximum flexibility, without reducing the quality of the donation.

The advent of oocyte and embryo vitrification has opened up new opportunities for reproductive scientists to improve the practice and results of IVF attempts. It is now established that vitrification of whole oocyte cohorts does not compromise, and may even improve, the results of IVF attempts. In addition, it is now clear that progesterone modulates the frequency of Gonadotropin-Releasing Hormone (GnRH) pulses and can strongly inhibit the pulsatile secretion of GnRH and LH and thereby inhibit the LH peak induced by increased plasma concentrations of GnRH and LH. estradiol. And, in the context of oocyte donation, the deleterious effects of ovarian stimulation on endometrial receptivity have no impact: the increase in progesterone levels during stimulation is not a concern in this group who will not benefit from an embryonic transfer.

Initially, progesterone stimulation protocols were performed during the luteal phase as part of the urgent preservation of fertility in cancer patients. The first European feasibility study was conducted and published in 2013 in normotensive patients. While the preliminary findings were not optimistic, many publications, from 2013, showed that this luteal strategy is effective without the addition of a GnRH antagonist, but imposes a freeze all strategy. In all these studies, whether it is luteal phase stimulation schemes, strategies of 2 consecutive stimulations, in the follicular and then luteal phase, or random-start stimulation protocol, the quality of the oocytes does not seem to be impacted, with identical implantation and birth rates in the control groups (conventional ovarian stimulation). The state of health of newborns and malformation rates are also identical to those of conventional protocols.

Although luteal phase endogenous progesterone levels appear to be sufficient to block the LH surge, recent publications have also shown the efficacy of exogenous progesterone, which can, without compromising the oocyte's competence, replace the use of an agonist or antagonist during the follicular phase. The advantages are oral administration and the reduction of potential costs, without any secondary effect on the competence of oocytes.

Different progestins were used. Kuang et al (2015) report the first randomized study studying an exogenous progestogen-based ovarian stimulation protocol using medroxyprogesterone acetate (MPA). Compared to a standard short protocol, with embryonic vitrification in both groups, the number of mature oocytes and the number of frozen embryos, the implantation and pregnancy rates after thawed embryo transfers were not significantly different. The same group published between 2015 and 2017, 4 studies validating micronized progesterone as an effective oral alternative to treatment with GnRH agonists for the prevention of premature LH surge during controlled ovarian stimulation for intracytoplasmic sperm injection (IVF-ICSI). Recently, the same group compared dydrogesterone and micronized progesterone with the same results. More recently, another progestogen, desogestrel, has been used in addition to corifollitropin alpha in an oocyte donation program, compared to a conventional antagonist protocol. The authors reported the same number of oocytes in both groups, with better tolerance of treatment in the desogestrel group. In the same way as for luteal phase stimulation protocols, exogenous progestin-exogenous ovarian stimulation protocols have similar neonatal outcomes, compared to "standard" protocols, for birth weight, gestational age, and Congenital malformation rate.

The use of luteal phase or follicular phase stimulation protocols with progestins could rapidly develop in the context of oocyte donation where no embryo transfer is performed. A single published study reports 13 MPA-blocked oocyte donor (PPO) cycles compared to counter-protocol donation cycles. This retrospective study found a significant difference in favor of the progestin-primed ovarian stimulation (PPOS) protocol for the number of oocytes retrieved. The duration of ovarian stimulation, the number of units of gonadotropins needed were not different from one group to another. No peak of LH was observed in the PPOS group.

These PPOS protocols have many advantages for these women wishing to donate their oocytes: improved flexibility (donors can choose the date of their oocyte retrieval, without cycle constraint), better acceptance with fewer injections, and lower cost. In addition, the use of Corifollitropin Alpha (CTA) improves patient comfort by reducing the number of injections (1 instead of 7), without altering the quality and number of oocytes. In addition, these protocols allow the initiation of ovulation by injection of GnRH agonists, drastically reducing the risk of hyperstimulation syndrome and contributing to the safety of donors. A retrospective study (proof of concept study) published in 2018 shows that the joint use of a PPOS and CTA gives satisfactory results, while being acceptable ("patient friendly").

To improve donor comfort and validate the use of progestogen-blocking ovarian stimulation protocols, this protocol combining the use of corifollitropin alpha and blocking the preterm-mediated progestogen LH peak is an innovative and promising approach, without impact neither on quantity nor on oocyte quality.

Our study (proof of concept) aims to validate the use of PPOS in oocyte donation, and to show that these stimulation protocols can be started whatever the phase of the menstrual cycle.

The assumptions are:

- The number of oocytes retrieved is not significantly different, regardless of the start date of treatment during the menstrual cycle.

Exogenous progestin therapy effectively blocks the LH surge during ovarian stimulation.

- It is possible to significantly reduce the number of injections during controlled ovarian stimulation for oocyte donors and the cost to society, without decreasing the effectiveness of ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Donor of oocytes having spontaneous and regular menstrual cycles, and having taken no hormonal treatment (in particular contraceptive) during the cycle preceding the donation.
* Patient with normal ovarian reserve with antral follicle count> 8,
* BMI between 18 and 32
* Regular natural menstrual cycles, and absence of hormonal treatment during the cycle preceding the donation cycle
* Major patient
* Affiliation to social security

Exclusion Criteria:

* Stage 3-4 endometriosis
* ovarian cyst> 30 mm,
* Polycystic ovary syndrome
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of oocytes punctured | 45 days
  Number of oocytes punctured after ovarian stimulation as described above, regardless of the phase of the menstrual cycle at the time of injection of corifollitropin alpha.

SECONDARY OUTCOMES:
Premature peak of LH | 45 days
  Frequency of occurrence of a premature peak of LH
Hyperstimulation syndrome | 45 days
  Occurrence of moderate to severe ovarian hyperstimulation syndrome
Number of injection | 45 days
  Number of injection is needed to evaluate the stimulation parameters
Number of Recombinant follicle stimulating hormone (r-FSH) units required for ovarian stimulation | 45 days
  the number of r-FSH units required for ovarian stimulation is needed to evaluate the stimulation parameters
Number of days of stimulation | 45 days
  The number of day of stimulation is needed to evaluate the stimulation parameters

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU Lille, Lille
  - CHU Bondy, Paris
  - CHU Tenon, Paris
  - Clinique de la Sagesse, Rennes

IPD SHARING:
Plan to Share IPD: No